CLINICAL TRIAL: NCT05139069
Title: Using Implementation Science to Increase Pre-Exposure Prophylaxis Uptake Among African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00012361
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Domestic Violence
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-Informed Pre-Exposure Prophylaxis Implementation Toolkit (Experimental): The Toolkit to be developed in the proposed study includes components from the women-specific Pre-Exposure Prophylaxis care continuum theoretical model and implementation challenges, and is adapted to identify and provide care to women experiencing intimate partner violence. Overall, the Toolkit is designed to create culturally-congruent, intimate partner violence-informed clinical settings; and equip clinical staff with the knowledge and skills they need to address HIV prevention for African American women; and integrate intimate partner violence into Pre-Exposure Prophylaxis care services.
  Interventions: Behavioral: Trauma-Informed Toolkit

INTERVENTIONS:
Behavioral: Trauma-Informed Toolkit — Staff in this intervention will be trained to conducting intimate partner violence screening, and providing support to women through referrals to local community resources; to help African American women identify and understand HIV risk factors (e.g., unprotected condom less sex with a male partner who is HIV-positive or unknown HIV status); and to communicate with their African American women patients in a respectful way in order to build trust and facilitate shared decision making.

SUMMARY:
Pre-exposure prophylaxis may be a viable option for African American women at-risk for HIV infection, but few studies have identified optimal strategies to reach African American women in need of Pre-Exposure Prophylaxis nor examined effective strategies to scale-up Pre-Exposure Prophylaxis among African American women in the South. African American women in the South experience high rates of intimate partner violence which could force women to choose between HIV prevention or intimate partner violence prevention. The proposed research study seeks to develop, pilot-test, and evaluate a Pre-Exposure Prophylaxis Implementation Toolkit within two community healthcare clinics located in Jackson, Mississippi to increase Pre-Exposure Prophylaxis uptake among African American, address intimate partner violence as a barrier to Pre-Exposure Prophylaxis uptake, and ultimately combat racial disparities in women's HIV diagnoses.

DETAILED DESCRIPTION:
HIV and intimate partner violence are intersecting, mutually-reinforcing epidemics that significantly affect African American women, particularly women in the U.S. South. African American women face some of the highest rates of both HIV and intimate partner violence among U.S. women, and these burdens are most pronounced in the South. African American surviving intimate partner violence may experience forced, condom less sex, which increases the risk of HIV acquisition. Pre-exposure prophylaxis has the potential to be the most innovative HIV prevention strategy, however it remains underutilized by African American women and residents of the South. In order to reduce African American women's HIV acquisition risk in the South, effective HIV prevention interventions need to concurrently address relationship safety and HIV acquisition risks. Developing effective interventions to tackle this HIV-related disparity among African American women is essential to reach national HIV goals.Therefore, the proposed research aims to develop, test, and evaluate a Pre-Exposure Prophylaxis Implementation Toolkit for clinical staff in community healthcare settings in the South. The Toolkit will be evaluated using the Reach, Effectiveness-Adoption, Implementation, Maintenance (RE-AIM). The Toolkit will serve the dual purpose of increasing Pre-Exposure Prophylaxis uptake among African American women in the South while addressing intimate partner violence as a potential Pre-Exposure Prophylaxis barrier. This research project will include a formative evaluation (i.e., reach stage), including key informant interviews with clinical staff at the partnering community healthcare clinics (N=10), and six focus groups with African American women at risk for HIV acquisition (i.e., Pre-Exposure Prophylaxis-eligible; %50 intimate partner violence-exposed). The qualitative data from the formal evaluation will inform the development of the Pre-Exposure Prophylaxis Implementation Toolkit, including detailed curriculum and supporting materials. The Toolkit will be pilot tested in two community healthcare clinics using a nonrandomized waitlist control design employed at the clinic-level. Clinic 1 will receive the Toolkit; and after the 8-month data is collected, Clinic 2 will receive the Toolkit. Changes in Pre-Exposure Prophylaxis uptake and retention in care will be assessed at the clinic level from 8-months before and after the Toolkit is implemented (i.e., effectiveness stage). To examine these effects at the clinic-level, a series of interrupted time series analyses will be conducted. This approach allows us to analyze population changes as opposed to individual change. To yield a moderate effect size with a power=.80 and alpha =.05, a sample size of at least 8 timepoints are needed. Following the Toolkit's implementation, four focus groups with clinical staff will be conducted to assess barriers and facilitators (i.e., adoption stage). Lastly, key informant interviews with clinical staff (N=20) will be conducted to assess fidelity of the Toolkit's components.

ELIGIBILITY:
Inclusion Criteria:

- currently providing care at a community healthcare clinic in Mississippi

Exclusion Criteria:

* non-English speaking
* inability to read and comprehend questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Clinic's proportion of women with Pre-Exposure Prophylaxis uptake | Baseline to 8-months after Toolkit implementation in each clinic
  Pre-Exposure Prophylaxis uptake will be classified as a woman receiving a Pre-Exposure Prophylaxis prescription from a pharmacy.
  Pre-Exposure Prophylaxis uptake will be coded as a binary variable (0=did not receive Pre-Exposure Prophylaxis prescription; 1=received Pre-Exposure Prophylaxis prescription) and will be obtained from clinic aggregated data.

SECONDARY OUTCOMES:
Clinic's proportion of women with Pre-Exposure Prophylaxis retention | Baseline to 8-months after Toolkit implementation in each clinic
  Pre-Exposure Prophylaxis retention will be classified as a woman attending scheduled three- and six-month followup visits. There will be a three and six-month follow-up visit variable and coded as binary (0=did not attend follow-up visit; 1= did attend follow-up visit).
Clinic's %Pre-Exposure Prophylaxis Uptake | Baseline to 8-months after Toolkit implementation in each clinic
  % Pre-Exposure Prophylaxis Uptake is calculated as the number of African American women who initiated Pre-Exposure Prophylaxis divided by the number of African American women who were offered Pre-Exposure Prophylaxis at the clinic.
Clinic's Pre-Exposure Prophylaxis Coverage | Baseline to 8-months after Toolkit implementation in each clinic
  % Pre-Exposure Prophylaxis Coverage will be calculated as the number of African American women using Pre-Exposure Prophylaxis divided by the number of African American women who visited the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Tiara C. Willie, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No